CLINICAL TRIAL: NCT04891614
Title: THE PRISM-PTSD PILOT TRIAL (Process-Instructed Self Neuro-Modulation ("Prism") Pilot Trial for Post-Traumatic Stress Disorder)
Brief Title: The PRISM Pilot Trial for Post-Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GrayMatters Health Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP001
Record Dates: First submitted 2021-05-06; First posted 2021-05-18 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-04

CONDITIONS: Post-Traumatic Stress Disorder (PTSD)
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: single-arm, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Subjects diagnosed with PTSD will be recruited from the community and from local clinical programs. All subjects will undergo Prism neurofeedback training.
  Interventions: Device: PRISM

INTERVENTIONS:
Device: PRISM — Subjects will complete 15 neurofeedback training sessions delivered twice per week, on non-consecutive days, over 8 consecutive weeks.

SUMMARY:
A Prospective, Single-Arm, Open-Label Pilot Trial, to Assess Safety and Effectiveness of Process-Instructed Self neuro-Modulation ("Prism"), as an Adjunct to Standard of Care, in Subjects with Post-Traumatic Stress Disorder (PTSD)

DETAILED DESCRIPTION:
Prism is a software device intended for neurofeedback (NF) training (i.e. operant condition based on EEG signals, also known as EEG-biofeedback), to be used in combination with a standard computer and supported EEG hardware. For purposes of this training, information for feedback is derived and processed from several EEG channels. Prism provides visual and/or auditory signals that correspond to the patient's computed EEG signal, which serves as a surrogate indicator of achieving a state of reduced amygdala activity.

The study is a Prospective, Single-Arm, Open-Label Pilot Trial, to Assess Safety and Effectiveness of Process-Instructed Self neuro-Modulation ("Prism"), as an Adjunct to Standard of Care, in Subjects with Post-Traumatic Stress Disorder (PTSD).

The study population will include subjects diagnosed with Post-Traumatic Stress Disorder (PTSD) from 1 year to 20 years after index trauma. The total expected enrollment is up to 100 subjects in one or more sites.

The study's primary objective is to assess the safety and effectiveness of fifteen (15) EEG-NF training sessions using the Prism software in reducing PTSD-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 22 to 65
2. Any gender
3. Diagnosis of PTSD, established according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V)
4. 1 to 20 years since index trauma
5. Ability to give signed, informed consent
6. Normal or corrected-to-normal vision
7. Normal or corrected to normal hearing
8. Subject is able to adhere to the study schedule

Exclusion Criteria:

1. Have completed two or more full courses of trauma-focused therapy in the past (i.e., EMDR, Prolong Exposure Therapy, etc.), eligibility will be deemed upon the clinical judgment of the investigator.
2. Lifetime diagnosis for schizophrenia, schizoaffective disorder, schizophreniform disorder, Bipolar I disorder, or delusional disorder
3. Any mood disorder and anxiety disorder according to DSM-5 (in addition to those described in Exclusion 2) that is the primary focus of treatment in the last 6 months prior to screening, as per the clinical judgment of the investigator
4. Lifetime diagnosis of autism, mental retardation at the discretion of the investigator.
5. Diagnosis of moderate or severe substance use disorder within the last 3 months of screening visit (as defined in DSM-5-substance use disorder) or at screening visit
6. Any prescribed Benzodiazepine which cannot be ceased for the duration of the study (with a washout period of at least 2 weeks prior to the first Prism training session) or which cannot be replaced with short-acting benzodiazepines that are taken only for sleeping during the night
7. Any psychotropic medication other than a stable dose of selective serotonin reuptake inhibitors (SSRIs) or serotonin-norepinephrine reuptake inhibitor (SNRIs)
8. Any change in or initiation of- SSRIs or SNRIs antidepressants within the past 4 weeks. At the time of recruitment, subjects must have no intention of changing their medication or psychotherapy during the study duration
9. Any suicidal behavior in the past 1 year (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior) prior to screening and during the screening period
10. Recent initiation (within the past 3 months) of cognitive-behavioral therapy or any evidence-based PTSD psychotherapy (Cognitive Processing Therapy [CPT], Prolonged Exposure [PE], Eye Movement Desensitization and Reprocessing [EMDR]); continuation of established maintenance supportive therapy will be permitted
11. Any history of brain surgery, of penetrating, neurovascular, infectious, or other major brain injury, of epilepsy, or of other major neurological abnormality (including a history of traumatic brain injury [TBI] with loss of consciousness for more than 24 hours or posttraumatic amnesia for more than 7 days)
12. Any unstable medical condition, as per the clinical judgement of the investigator
13. In process of establishing/changing governmental/institutional compensation payments for PTSD symptoms
14. Enrollment in another clinical study at screening or within 2 months prior to screening, or intended enrollment within the duration of this study
15. Women who are pregnant, nursing, or who plan to become pregnant while in the trial

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-11-29 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS - 5) | Baseline visit (Week 1) and 3 month Follow-up visit
  The primary objective of this study is to assess the proportion of subjects who demonstrate clinically meaningful improvement in the Clinician Administered PTSD Scale (CAPS - 5) score from Baseline to the 3 months follow-up visit. Clinically meaningful improvement is defined here as a 6-point reduction or more in the CAPS-5 score.

SECONDARY OUTCOMES:
PCL-5 response rate | Baseline visit (Week 1), Post-Intervention Visit (Week 9) and 3 month Follow-up visit
  To assess the proportion of subjects who demonstrate clinically meaningful improvement in the PTSD Checklist for DSM-5 (PCL-5). Clinically meaningful improvement is defined here as a 10-point reduction or more in the PCL-5 score
ERQ score | Baseline visit (Week 1), Post-Intervention Visit (Week 9) and 3 month Follow-up visit
  Change from baseline to Month 3 visit in ERQ score
PHQ-9 score | Baseline visit (Week 1), Post-Intervention Visit (Week 9) and 3 month Follow-up visit
  Change from baseline to Month 3 visit in PHQ-9 score
Clinical Global Impression (CGI) | Baseline visit (Week 1), Post-Intervention Visit (Week 9) and 3 month Follow-up visit
  Change from baseline to Month 3 visit in CGI score

OTHER OUTCOMES:
Abbreviated PCL (APCL) | through study completion, an average of 8 weeks
  To assess the change in the score of the abbreviated PCL scale (APCL, assessed weekly during the EFP-NF training period)
learning success of the EFP-based neurofeedback | through study completion, an average of 8 weeks
  To quantify the learning success of the EFP-based neurofeedback (namely: learning volitional down-regulation of the Amyg-EFP signal, over time, during the EFP-NF training period)
Patient satisfaction survey | through study completion, an average of 5 month
  To quantify patient satisfaction from the EFP-NF training using survey
Remission rate | Baseline visit (Week 1), Post-Intervention Visit (Week 9) and 3 month Follow-up visit
  To assess the Remission rate at post training visit (8-9 weeks) and at the 3 months follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Adar Shani, Study Director — GrayMatters Health
Locations (5):
- NYU Langone Health, New York, New York, United States
- Israel (4):
  - Barzilai Medical Center, Ashkelon
  - Rambam Health Care Campus, Haifa
  - Mental Health Center in Be'er Ya'akov, Ness Ziona
  - Sheba Medical Center, Ramat Gan

IPD SHARING:
Plan to Share IPD: No